CLINICAL TRIAL: NCT04363047
Title: Immune Cells and the Coronavirus for Inflammatory Arthritis
Brief Title: Immune Cells in Inflammatory Arthritis With Coronaviruses, Including COVID-19
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr. Sebastien Viatte, Lecturer in Genetics, University of Manchester
Other Study IDs: 282566
Record Dates: First submitted 2020-04-20; First posted 2020-04-27 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: SARS Virus
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Volunteers: These people will have already provided at least one sample as part of the National Repository Healthy Volunteer Study.
  We aim to take blood samples from participants who have recovered from COVID-19 and compare them with blood samples we already have which were taken before the COVID-19 pandemic.
  We will need to compare these samples to other samples, so we will also need to blood samples from people who have not had COVID-19 (who have either tested negative or never had any symptoms).
  Interventions: Other: 40ml blood sample
- Rheumatoid Arthritis: These people will have already provided at least one sample as part of the BRAGGSS Study.
  We aim to take blood samples from participants who have recovered from COVID-19 and compare them with blood samples we already have which were taken before the COVID-19 pandemic.
  We will need to compare these samples to other samples, so we will also need to blood samples from people who have not had COVID-19 (who have either tested negative or never had any symptoms).
  Interventions: Other: 40ml blood sample

INTERVENTIONS:
Other: 40ml blood sample — We'll be collecting cells, DNA and serum.

SUMMARY:
A team at the University of Manchester are developing a test that tcould be helpful in detecting immunity to the Coronavirus (which causes the COVID-19 disease) in participants with inflammatory arthritis. It is based on a flu assay has already developed; the team will replace the flu antigen with a Coronavirus antigen to see if it is effective.

This project aims to develop a test to see if people who have had the virus have developed immunity to it. This could help to predict who might or might not get the disease a second time, who should stay at home to be protected from potential infection or who will not develop any symptoms, even if exposed to the virus.

When vaccination trials against the Coronavirus will be launched, this test could also help to see if the vaccine is effective.

ELIGIBILITY:
Inclusion Criteria:

* Has previously taken part in either the BRAGGSS or National Repository Healthy Volunteer Study
* Has agreed to be contacted abut future research projects
* Has previously provided a blood sample for either the BRAGGSS or National Repository Healthy Volunteer Study
* Is willing to complete the informed consent form, registration slip, questionnaire and provide a 40ml blood sample
* Has a good written understanding of English

Exclusion Criteria:

* Has not previously taken part in either the BRAGGSS or National Repository Healthy Volunteer Study
* Has not agreed to be contacted abut future research projects
* Has not previously provided a blood sample for either the BRAGGSS or National Repository Healthy Volunteer Study
* Is not willing to complete the informed consent form, registration slip, questionnaire and provide a 40ml blood sample
* Has not got a good written understanding of English

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: People who have previously taken part in (and provided at least 1 set of blood samples to) either the BRAGGSS or National Repository Healthy Volunteer Studies and have given us permission to contact them for future research
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence and abundance of CD4+ T lymphocytes | 2 years
  the prevalence and abundance of CD4+ T lymphocytes specifically recognizing SARS-CoV-2 in COVID-19 patients with inflammatory arthritis, in pre- and post-infection samples; in patients without COVID-19 and in healthy volunteers with or without COVID-19. Correlation of these cells with COVID-19 severity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No